CLINICAL TRIAL: NCT00657423
Title: Study of Endostar Combined With Docetaxel and Cisplatin on the Angiogenesis of Advanced Non-small Cell Lung Cancer
Brief Title: Impact of Endostar Combined With Chemotherapy on the Angiogenesis of Advanced Non-small Cell Lung Cancer (NSCLC)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Yantai Medgenn Ltd. (Industry)
Responsible Party: Shengqing Li, Dept.of Respiratory Diseases, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: XJ-EnXS0802
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2010-09-17 (Estimated); Status verified 2008-08

CONDITIONS: Lung Neoplasms
Keywords: Lung Neoplasms; Endostatins; Vascular Endothelial Growth Factors; Fibroblast Growth Factors; Survival Rate
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Cisplatin; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Treated by endostar combined with docetaxel and cisplatin
- 2 (Active Comparator)
  Interventions: Drug: Treated by docetaxel and cisplatin

INTERVENTIONS:
Drug: Treated by endostar combined with docetaxel and cisplatin — recombinant human endostatin given intravenously,7.5mg/㎡,d1-14,2cycles. docetaxel given intravenously,75mg/㎡,d1,2cycles. cisplatin given intravenously,75mg/㎡,d1,2cycles.
  Other Names: Endostar; Taxotere
  Arms: 1
Drug: Treated by docetaxel and cisplatin — docetaxel given intravenously,75mg/㎡,d1,2cycles. cisplatin given intravenously,75mg/㎡,d1,2cycles.
  Other Names: Taxotere
  Arms: 2

SUMMARY:
To study the impact of endostar combined with docetaxel and cisplatin on the angiogenesis of non-small cell lung cancer, patients will be randomly assigned to the group one (endostar combined with docetaxel and cisplatin) and group two (docetaxel and cisplatin).

* The serum concentrations of Endostatin,VEGF and bFGF are determined.
* Blood circulating endothelial cells (CECs) and circulating hematopoietic progenitor cells (CPCs) will be measured by flow cytometer.
* Statistical analysis will be applied to study the relationship between the levels of Endostatin, VEGF, bFGF, CECs and CPCs and the clinical outcomes such as objective response rate(ORT), time to progression (TTP), mean survival time(MST), toxicity and quality of life (QOL).

DETAILED DESCRIPTION:
To study the impact of endostar combined with docetaxel and cisplatin on the angiogenesis of non-small cell lung cancer,patients will be randomly assigned to the experimental group(endostar combined with docetaxel and cisplatin) and the control group (docetaxel and cisplatin).

* the serum concentrations of Endostatin,VEGF and bFGF are determined.
* Blood circulating endothelial cells (CECs) and circulating hematopoietic progenitor cells (CPCs) will be measured by flow cytometer.
* the clinical parameters such as objective response rate (ORT),time to progression(TTP) and mean survival time(MST) will be collected according to the WHO criteria.
* the toxicity will be recorded according to the NCI-CTC v3.0.
* the Quality of life was self-assessed using the European Organisation for Research and Treatment of Cancer (EORTC) QLQ C-30 questionnaire.
* Statistical analysis will be applied to study the relationship between the levels of Endostatin,VEGF,bFGF,CECs and CPCs and the clinical outcomes such as ORT, TTP, MST, toxicity and QOL.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of advanced or metastatic NSCLC (confirmed histologically, with a tumor that was measurable by clinical and/or radiologic examination.
* Have an Eastern Cooperative Oncology Group performance status 0 to 2.
* Adequate renal, cardiac, hepatic, and hematologic function as indicated by the following parameters: absolute neutrophil count 2 x the ninth power of ten/L, thrombocytes 100 x the ninth power of ten/L, hemoglobin 10 g/dL, total bilirubin 1.25x the upper limit of normal range (ULN), ALT and AST 1.5x ULN, alkaline phosphatase 5x ULN, creatinine 1.15x ULN.

Exclusion Criteria:

* Known brain metastases or secondary neoplasia.
* Myocardial insufficiency or myocardial infarction within the preceding 6 months.
* Severe renal or hepatic insufficiency.
* Pre-existing motor or sensor neurotoxicity WHO grade 2.
* Severe psychologic disease.
* Active infection, or other condition that could compromise protocol compliance.
* Simultaneous administration of other antineoplastic medications.
* Clinically significant hemoptysis.
* Pregnancy and/or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-12 (Estimated); Study Completion 2009-04 (Estimated)

PRIMARY OUTCOMES:
mean survival time | 1 year

SECONDARY OUTCOMES:
objective response rate | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Changgui Wu, MD, PHD, Principal Investigator — Dept. Resp. Diseases, Xijing Hospital
Locations (1):
- Dept. Resp. Diseases, Xijing Hospital, Xi'an, Shaanxi, China